CLINICAL TRIAL: NCT02119273
Title: Systemic Corticosteroids in the Perioperative Management of Chronic Rhinosinusitis Without Nasal Polyps (CRSsNP)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Kristin Seiberling, MD, Physician, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5140031
Record Dates: First submitted 2014-03-20; First posted 2014-04-21 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Chronic Rhinosinusitis Without Nasal Polyps (CRSsNP)
Keywords: CRSsNP; Steroids; Corticosteroids; Endoscopic; Surgery; Perioperative
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Steroid (Experimental): The steroid arm will take prednisone 10mg tabs starting 7 days prior to surgery with a taper (4 tabs/day for 3 days, 3 tabs/day for 3 days, 2 tabs/day for 3 days, 1 tab/day for 3 days).
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator): The placebo arm will receive placebo pills identical in appearance to prednisone 10mg pills. They will start taking them 7 days prior to surgery with a taper (4 tabs/day for 3 days, 3 tabs/day for 3 days, 2 tabs/day for 3 days, 1 tab/day for 3 days).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — See arm description
  Arms: Steroid
Drug: Placebo — See arm description
  Arms: Placebo

SUMMARY:
Oral corticosteroids are commonly utilized for the management of chronic rhinosinusitis with and without nasal polyps (CRSwNP and CRSsNP, respectively). Although strong evidence supports the benefit of routine and perioperative oral corticosteroids for CRSwNP, there is limited evidence to support their utility for CRSsNP. The investigators intend to perform a randomized, double blind, placebo controlled clinical trial to investigate the impact of steroids used within 2 weeks prior to surgery for CRSsNP. Patients with CRSsNP that present to the investigators office will be included if they have failed maximal medical management and have elected to undergo endoscopic sinus surgery (ESS) after July 1, 2014. The investigators hypothesis is that oral corticosteroids given 2 weeks prior to surgery will improve subjective and objective outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (ages 18-80) with a diagnosis of chronic rhinosinusitis without nasal polyps (CRSsNP) that have failed a 6 week trial of maximal medical therapy and have elected to undergo endoscopic sinus surgery will be offered enrollment in this study.
* Diagnosis of chronic rhinosinusitis (CRS) is based on the European Position on Rhinosinusitis (EPOS) 2012 guidelines.
* These include a greater than 12 week history of inflammation of the nose or paranasal sinuses characterized by at least 2 symptoms.
* These symptoms must include at least one of the following:

  * nasal obstruction
  * rhinorrhea
  * postnasal drip.
* Additional symptoms can include facial pain/pressure or anosmia/hyposmia.
* These symptoms must be supplemented by either endoscopic signs of disease or characteristic CT changes.
* The presence or absence of nasal polyps defines the subtype (with polyps: CRSwNP; without polyps: CRSsNP).

Exclusion Criteria:

* Patients will be excluded if they have nasal polyps or suspected allergic fungal rhinosinusitis (AFRS) based on classic endoscopy and CT findings.
* Additionally, patients with known immunocompromise or mucociliary disorders will be excluded.
* Patients that received oral corticosteroids within 6 weeks prior to the planned surgery will also be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Lund-Kennedy Endoscopy Score (LKES) | 12 weeks
  Objective endoscopic measure of sino-nasal mucosal health

SECONDARY OUTCOMES:
Sino-nasal Outcomes Test (SNOT-22) | 12 weeks
  Patient completed survey that objectifies sinonasal symptoms
Boezaart bleeding score | Day of surgery
  Surgeon completed survey of bleeding during surgery
Estimated blood loss | Day of surgery
  Estimation of blood lost during surgery, as reported by anesthesiologist
Difficulty of surgery score | Day of surgery
  Surgeon completed survey of surgical difficulty

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Seiberling, MD, Principal Investigator — Loma Linda Department of Otolaryngology
Locations (1):
- Loma Linda Sinus and Allergy Center, Redlands, California, United States